CLINICAL TRIAL: NCT05543837
Title: Effect of Capsaicin on the Augmentation of Cerebral Perfusion. A Phase II Study.
Brief Title: Capsaicin for Cerebral Perfusion Augmentation
Acronym: CCPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Centenario Hospital Miguel Hidalgo (Other)
Responsible Party: Principal Investigator, Juan Manuel Marquez Romero, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-E-20
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Circulatory Disorder
Keywords: capsaicin; cerebal perfusion
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capsaicin .66μMol/ml (Experimental): Group receiving .66μMol/ml
  Interventions: Drug: Capsaicin
- Capsaicin .99μMol/ml (Experimental): Group receiving .99μMol/ml
  Interventions: Drug: Capsaicin

INTERVENTIONS:
Drug: Capsaicin — Patients will receive a fixed dose of capsaicin
  Other Names: 8-Methyl-N-vanillyl-trans-6-nonenamide

SUMMARY:
To determine the effect of capsaicin upon serial transcranial Doppler (TCD) markers of cerebral blood flow (CBF). Methods Serial TCD testing in 30 participants with cerebrovascular risk factors. Capsaicin doses .66 and .99 μMol. Outcomes: peak systolic and end-diastolic velocities in the middle cerebral artery (MCA), mean velocity (MV), pulsatility index (PI), CBF index, arterial pressure, and perceived pungency (PP) in five minutes intervals up to 20 minutes.

DETAILED DESCRIPTION:
Subjects The study is expected to enroll 30 participants who will be recruited from the Internal Medicine outpatient clinic. Those willing to participate will be asked to sign the informed consent form (ICF) and will received the assigned dose of capsaicin. Half of the participants in each dose group will receive stimulation on either left or right side of the palate, but TCD measurements will be bilateral. Chemical stimuli From an initial 0.1% capsaicin (Sigma-Aldrich, St. Louis, MO) stock solution in 95% ethanol; solutions with 66 and 99 μMol/ml solutions will be obtained by diluting the stock solution with distilled water. One milliliter of each dilution was pipetted on to 2 cm filter paper squares. Then, the filter papers will be let dry. Immediately before application, filter papers will be rehydrated with 1 milliliter of distilled water. The rehydrated filter paper will be applied and will remain stationary on the subject's hemi palate's posterior surface during TCD measurements. Participants will be instructed not to swallow and to avoid touching the paper filter with their tongue for the 20 minutes of the experiment.

TCD testing With a TCD device (Philips Sonos 7500®) will include: peak systolic velocity (PSV) and end-diastolic velocity (EDV) in the middle cerebral artery (MCA) through the temporal window of the stimulated side. After a basal recording post stimulation recordings will initiate immediately after stimulation, and will be followed by serial recordings every five minutes and up to 20 minutes. At each time point the systolic pressure (SP), diastolic pressure (DP), and perceived pungency (PP) on a visual analog scale will be recorded. TCD markers of cerebral blood flow From the initial measurements the Mean velocity (MV) = EDV + [(PSVEDV) / 3], pulsatility index (PI) = PSV - EDV / MV, mean arterial pressure (MAP) = ((2 * DP) + SP) / 3 and, the CBF index (CBFi), CBFi = (MAP * 10) / 1.47^PI, will be calculated.

Statistical analysis Shapiro Wilkins W-Test for normality. The results of the continuous variables will be described as median (max-min) or mean+/- SD according to distribuition. The categorical variables will be described as tables of absolute and relative frequencies, and the comparisons between the groups of subjects (according to the dose of capsaicin) will be carried out with chi-square tests. To compare the variables studied between the groups of subjects (according to the different doses of capsaicin), Mann-Whitney U-Test/independent samples Student´s T-Test will be used appropriately. For comparisons of the baseline state with the changes recorded over time, various Wilcoxon signed-rank tests will be performed.The relationship between pungency ratings and MV response will be evaluated by Spearman's rho test. The level of statistical significance will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Previous diagnosis and stable condition of one of the following:

Diabetes Mellitus Hypertension Dyslipidemia Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

* History of alergy or hypersensibility to dietary capsaicin
* Previous diagnosis of stroke
* Chronic use of cholinergic/anticholinergic drugs
* Chronic use of sympathomimetic drugs
* Chronic use of serotonergic drugs
* Chronic use of dopaminergic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Mean velocity | 20 minutes
  The Mean velocity in the Middle Cerebral Artery
Pulsatility Index | 20 minutes
  A calculated flow parameter in ultrasound, derived from the maximum, minimum, and mean Doppler frequency shifts during a defined cardiac cycle.

SECONDARY OUTCOMES:
Mean arterial pressure (MAP) | 20 minutes
  The average arterial pressure throughout one cardiac cycle, systole, and diastole.
Cerebral Blood Flow index | 20 minutes
  The result of the following formula: CBFi = (MAP * 10) / 1.47^Pulsatility Index.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Marquez-Romero, MD, MSc, Principal Investigator — Unidad de Medicina de Alta Especialidad, Torre Medica CMQ
Locations (1):
- Centenario Hospital Miguel Hidalgo, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with any qualified investigator upon request to the PI after signing a data use agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months
Access Criteria: Any qualified investigator in the field